CLINICAL TRIAL: NCT02527512
Title: Bacterial Wound Contamination Prior to Closure: Povidone-Iodine Versus Saline Irrigation in Pediatric Spine Fusion Surgery
Brief Title: Bacterial Contamination: Iodine vs Saline Irrigation in Pediatric Spine Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Michael Glotzbecker, Assistant Professor, Orthopaedic Surgery, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-P00015085
Record Dates: First submitted 2015-08-07; First posted 2015-08-19 (Estimated); Results first posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-04

CONDITIONS: Surgical Site Infection
Keywords: Scoliosis; Spine fusion; 0.35% povidone-iodine
MeSH Terms: conditions — Surgical Wound Infection; Scoliosis | interventions — Povidone-Iodine; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Povidone-Iodine (Active Comparator): 0.35% povidone-iodine ("Betadine")
  Interventions: Drug: Povidone-Iodine
- Normal Saline (Active Comparator): Sterile sodium chloride (NaCl) solution
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Povidone-Iodine — Chemical complex of polyvinylpyrrolidone (povidone, PVP) and elemental iodine
  Other Names: Betadine
  Arms: Povidone-Iodine
Other: Normal Saline — Solution of 0.90% w/v of NaCl, 308 mOsm/L or 9.0 g per liter
  Other Names: NSS, NS or N/S
  Arms: Normal Saline

SUMMARY:
This study will evaluate the safety of povidone-iodine irrigation in pediatric spinal patients by collecting pre- and post-operative safety labwork. Furthermore, the efficacy of povidone-iodine and normal saline irrigation at reducing bacterial contamination of the surgical wound will be measured by collecting cultures before and after irrigation.

DETAILED DESCRIPTION:
Previous research has shown there is baseline bacterial contamination of surgical spinal wounds prior to closure. While this bacterial contamination may or may not lead to infection, recent adult studies demonstrated reduced infection rates by using povidone-iodine irrigation before closure. This study will determine the safety of using povidone-iodine irrigation in pediatric spinal patients and how effective it is at reducing bacterial contamination of the spinal surgical wound prior to closure, compared with normal saline. The investigators hypothesize povidone-iodine is both safe and effective. Understanding techniques that reduce the local bacterial load in the wound prior to closure after spinal fusion will give data to support measures that will ultimately reduce the rate of postoperative infections.

ELIGIBILITY:
Inclusion Criteria:

1. Age 3 to 18 years on day of surgery
2. diagnosis of spinal deformity
3. undergoing elective posterior spine multi-level instrumentation surgery

Exclusion Criteria:

1. Documented renal failure
2. documented allergy to iodine or shellfish
3. previous spine fusion surgery
4. undergoing elective posterior spine single-level instrumentation surgery
5. undergoing anterior spine multi-level instrumentation surgery
6. current antibiotic use.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 173 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Glotzbecker, MD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Children's Mercy Kansas City, Kansas City, Missouri
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dietz FR, Koontz FP, Found EM, Marsh JL. The importance of positive bacterial cultures of specimens obtained during clean orthopaedic operations. J Bone Joint Surg Am. 1991 Sep;73(8):1200-7. PMID 1890121
- [Background] Nandyala SV, Schwend RM. Prevalence of intraoperative tissue bacterial contamination in posterior pediatric spinal deformity surgery. Spine (Phila Pa 1976). 2013 Apr 15;38(8):E482-6. doi: 10.1097/BRS.0b013e3182893be1. PMID 23370682
- [Background] Chang FY, Chang MC, Wang ST, Yu WK, Liu CL, Chen TH. Can povidone-iodine solution be used safely in a spinal surgery? Eur Spine J. 2006 Jun;15(6):1005-14. doi: 10.1007/s00586-005-0975-6. Epub 2005 Aug 20. PMID 16133077
- [Background] Cheng MT, Chang MC, Wang ST, Yu WK, Liu CL, Chen TH. Efficacy of dilute betadine solution irrigation in the prevention of postoperative infection of spinal surgery. Spine (Phila Pa 1976). 2005 Aug 1;30(15):1689-93. doi: 10.1097/01.brs.0000171907.60775.85. PMID 16094267

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 6 patients that were ineligible after enrollment and were excluded prior to group assignment. The reasons included: fused fewer levels than planned(< 6 levels), surgeon forgot to take swap samples, excessive bleeding and transfusion, put on antibiotic after enrollment and one family asked to be removed after enrollment. Thus, a total of 167 subjects were assigned to treatment groups.
Period: Overall Study
Arm/Group | Povidone-Iodine | Normal Saline
Started | 85 | 82
Completed | 77 | 76
Not Completed | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Povidone-Iodine | Normal Saline | Total
Number analyzed (Participants) | 77 | 76 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (2.39) | 14.8 (2.04) | 14.7 (2.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 60 | 122
  Male | 15 | 16 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 59 | 49 | 108
  Race: Black/ African American | 4 | 5 | 9
  Race: Asian | 1 | 2 | 3
  Race: American Indian/ Alakan Naitive | 0 | 0 | 0
  Race: Native Hawaiian/ Pacific Islander | 0 | 0 | 0
  Race: Unknown/ Refused/ Missing | 13 | 20 | 33
ASA [Count of Participants; unit: Participants] — The American Society of Anesthesiologists' Classiﬁcation of Physical Health Classification was used to asses perioperative risks and patients that were classified as ASA I-IV were included for the study:
  ASA I- A normal healthy person ASA II- Mild systemic diseases ASA III- Severe systemic disease with substantive functional limitations ASA IV- Severe systemic disease that is a constant threat to life
  ASA I group is predictive of better outcomes while ASA IV is associated with least favorable treatment outcome.
  Participants
    1 | 23 | 20 | 43
    2 | 34 | 34 | 68
    3 | 19 | 22 | 41
    4 | 1 | 0 | 1
Risk Group [Count of Participants; unit: Participants]
  Low risk (idiopathic) | 59 | 57 | 116
  High risk (other etiologies) | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Culture Positivity
Description: Assess feasibility of a larger randomized controlled trial using significance of differences in the bacteriology and contamination rates of both treatment arms. Also measured baseline tissue colonization rates.
Time Frame: Cultures taken before and after irrigation during surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Povidone-Iodine | Normal Saline
Number analyzed (Participants) | 77 | 76
Participants
  pre-washout: bacteria present | 14 | 13
  pre-washout: bacteria absent | 63 | 63
  post-washout: bacteria present | 12 | 14
  post-washout: bacteria absent | 65 | 62

2. Secondary Outcome: Risk Groups
Description: Baseline (pre-irrigation) and post-irrigation tissue colonization rates and changes in culture positivity
Time Frame: Cultures taken before and after irrigation during surgery
Measure: Count of Participants; unit: Participants
Groups:
- High Risk Povidone-iodine; High Risk Saline: congenital, neuromuscular, and syndromic deformities
- Low Risk Povidone-iodine; Low Risk Saline: idiopathic deformities
Arm/Group | High Risk Povidone-iodine | High Risk Saline | Low Risk Povidone-iodine | Low Risk Saline
Number analyzed (Participants) | 18 | 19 | 59 | 57
Participants
  pre-irrigation: positive | 2 | 3 | 12 | 10
  pre-irrigation: negative | 16 | 16 | 47 | 47
  post-irrigation: positive | 5 | 4 | 7 | 10
  post-irrigation: negative | 13 | 15 | 52 | 47

ADVERSE EVENTS:
Time Frame: Up to 90 days postoperatively
Arm/Group | Povidone-Iodine | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/76
Other Adverse Events (participants affected / at risk) | 0/77 | 0/76

LIMITATIONS AND CAVEATS:
While this study was underpowered to detect a statistically significant difference between the study arms, a difference may not exist. If a difference does exist, it would require a large cohort to be statistically significant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT02527512/Prot_SAP_002.pdf
  • Informed Consent Form (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/12/NCT02527512/ICF_003.pdf